CLINICAL TRIAL: NCT02204202
Title: Positron Emission Tomography Assessment of Acute Lung Transplant Rejection
Brief Title: PET Assessment of Acute Lung Transplant Rejection
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01HL121218-01-201102155; R01HL121218 (NIH)
Record Dates: First submitted 2014-07-24; First posted 2014-07-30 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Lung Disease
Keywords: acute lung transplant rejection; neutrophilic lung inflammation; positron emission tomography imaging; [18F] fluorodeoxyglucose; [18F] ISO-1
MeSH Terms: conditions — Lung Diseases | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — cells from bronchoalveolar lavage specimen; tissues from biopsy specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Grade A0: Double-lung transplant recipients with no evidence of rejection who undergo both [18F]FDG and [18F]ISO-1 PET imaging scans
  Interventions: Drug: [18F]FDG; Drug: [18F]ISO-1
- Grades A2-3: Double-lung transplant recipients with mild to moderate rejection who undergo both [18F]FDG and [18F]ISO-1 PET imaging scans
  Interventions: Drug: [18F]FDG; Drug: [18F]ISO-1

INTERVENTIONS:
Drug: [18F]FDG — 10 millicuries (mCi) of [18F]FDG will be injected intravenously at the start of a 60-minute dynamic PET scan acquisition
  Other Names: fluorodeoxyglucose
Drug: [18F]ISO-1 — 8 mCi of [18F]ISO-1 will be injected intravenously at the start of a 60-minute dynamic PET scan acquisition
  Other Names: F-18 labeled proliferation tracer targeting PGRMC1

SUMMARY:
The purpose of this research study is to gain understanding of the basic responses of the lungs to inflammation and specifically if there may be a better way to detect graft inflammation using non-invasive methods as well as to determine the effectiveness of immunosuppressive treatment regimens in preventing acute rejection in lung transplant recipients.

DETAILED DESCRIPTION:
Positron emission tomography with fluorodeoxyglucose (FDG-PET) is a potential way we can measure lung inflammation. FDG-PET imaging is a clinically accepted and FDA-approved method that is commonly used in the diagnosis and management of cancer. PET is a machine that detects radiation and generates pictures using a donut shaped scanner similar in appearance to an x-ray "CAT" computerized axial tomography or computed tomography (CT) scan. FDG stands for [18F] (flourine 18) fluorodeoxyglucose, a radiolabeled sugar that is used to identify areas of inflammation with the PET scanner. A CT scan takes a picture of what the lungs and airways look like.

T cells are the primary cause of acute rejection of lung transplants. Because T cells must divide in order to be activated and cause rejection, imaging them while they are dividing is another way that we can determine whether acute rejection is occurring. A new PET tracer called [18F]ISO-1 (18F-labeled σ2-receptor ligand for PET, N-(4-(6,7-dimethoxy-3,-4-dihydroisoquinolin-2(1H)-yl)butyl)-2-(2-18F-fluoroethoxy)-5-methylbenzamide (18F-3c), binds to dividing cells. Therefore, [18F]ISO-1 may help us measure acute rejection more accurately. [18F]ISO-1 is an investigational drug.

ELIGIBILITY:
Inclusion Criteria:

* Double-lung transplant recipient
* Scheduled for bronchoscopy with transbronchial biopsy
* Capable of lying still and supine with arms raised above the head within the PET/CT scanner for ~1.25 hours
* Capable of following instructions for breathing protocol during CT portion of PET/CT
* Able and willing to give informed consent
* BMI < 35
* Already scheduled to undergo bronchoscopy with bronchoalveolar lavage (BAL) for clinical reasons
* Willing to donate a portion of BAL and biopsy specimen for laboratory testing

Exclusion Criteria:

* Glucose level > 150 mg/dl at time of [18F]FDG PET scan (however, up to 160 mg/dl, with repeat testing showing level is stable or decreasing, is acceptable)
* Pregnancy (confirmed by qualitative urine human chorionic gonadotropin (hCG) pregnancy test)
* Lactation
* Presence of implanted electronic medical device
* Enrollment in another research study of an investigational drug
* Inability to lie flat with arms raised above the head for 1.5 hours for PET/CT scans or follow breathing protocol instructions for the CT portion of the PET/CT

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient within 7 months of double-lung transplantation and who is scheduled for bronchoscopy with biopsy will be eligible. Patients will be identified via the bronchoscopy schedule through the Lung Transplant Center at Barnes-Jewish Hospital / Washington University School of Medicine and approached for potential participation prior to their scheduled bronchoscopy. PET/CT imaging with [18F]FDG will be performed, if consented, no more than 3 days after results from the biopsy are reported. [18F]ISO-1 PET/CT imaging will be performed the day after [18F]FDG PET and can be performed after treatment for acute rejection has been initiated. We intend to image 30 lung transplant recipients with no evidence of rejection (grade A0) and 30 recipients with mild to moderate (grades A2-3) rejection.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2017-02-04 (Actual); Study Completion 2017-02-04 (Actual)

PRIMARY OUTCOMES:
Ki, the influx constant that describes the rate of [18F]FDG uptake, in the whole lung | This outcome measure is assessed from the [18F]FDG scan performed on Day 1.
Logan plot analysis determined distribution volume ratio (DVR) of [18F] ISO-1 uptake | This outcome measure is assessed from the [18F]ISO-1 PET scan performed on Day 2.

SECONDARY OUTCOMES:
Progesterone receptor membrane component 1 (PGRMC1) staining of biopsy tissues and bronchoalveolar lavage cells | Assessed after the baseline clinical bronchoscopy procedure is performed 3 days prior to FDG PET/CT scan
  The biopsy specimens will be stained for proliferation markers. The bronchoalveolar lavage cells will be assessed for glucose uptake with 2-NBDG ( fluorescent glucose analog that has been used to monitor glucose uptake in live cells, as an indicator of cell viability).

CONTACTS AND LOCATIONS:
Overall Officials: Delphine L Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine / Barnes-Jewish Hospital, St Louis, Missouri, United States